CLINICAL TRIAL: NCT02513901
Title: Safety and Efficacy of the Histone Deacetylase Inhibitor Chidamide in Combination With Antiretroviral Therapy for Eradication of the Latent HIV-1 Reservoir(CHARTER)
Brief Title: Chidamide in Combination With Antiretroviral Therapy for Eradication of the Latent HIV-1 Reservoir
Acronym: CHARTER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Principal Investigator, Yongtao Sun, MD, PhD, Director of Department of Infectious Diseases, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015TD-Chidamide
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic HIV Infections
Keywords: Chidamide; Histone Deacetylase Inhibitor; HIV-1 Reservoir; Chronic HIV infections; Antiretroviral Therapy; HIV Eradication
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide (Experimental): Step 1 - Six participants will receive Chidamide 10 mg twice a week(BIW) for 4 consecutive weeks.
  Step 2 - Another six participants will receive Chidamide 30 mg twice a week(BIW) for 4 consecutive weeks.
  Participants will be enrolled into Step 1 first; if the dose given to Step 1 is well tolerated and no safety concerns are noted, Step 2 will be enrolled.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide will be given by mouth on Day 0, 3, 7, 10, 14, 17, 21, 24.
  Other Names: CS055; HBI-8000

SUMMARY:
HIV replication can be effectively suppressed and acquired immunodeficiency syndrome(AIDS) can be prevented with highly active antiretroviral therapy (HAART). However, HIV-infected people must remain on treatment continuously to avoid viral rebound and progression to AIDS. HIV persistence is thought to stem primarily from the presence of integrated copies of the proviral genome within long-lived cells. Because active viral gene expression causes cell death due to viral cytopathic effects and the immune response, long-lived cells likely harbor transcriptionally silent, latent provirus. HIV-1 persistence in long-lived cellular reservoirs remains a major barrier to a cure. HDACi have the potential to activate ("Kick") these latently infected cells. This will make the HIV infected cells visible to the immune system; the immune response and antiretrovirals(ARVs) will be able to attack and eliminate ("Kill") the infected cells. The purpose of this study is to evaluate the safety and efficacy of multi-dose Chidamide in combination with antiretroviral therapy in HIV-infected adults with suppressed viral load.

DETAILED DESCRIPTION:
Every participant will receive oral Chidamide on Day 0, 3, 7, 10, 14, 17, 21, 24. In Step 1, the dose of Chidamide will be 10 mg each time, for Step 2 30 mg each time. Participants will be enrolled into Step 1 first; if the dose given to Step 1 is well tolerated and no safety concerns are noted, Step 2 will be enrolled. All participants will keep their antiretroviral therapy during this study.

Each step of this study will last for 56 days, involving 14 study visits(Screening, Day 0, 2, 3, 8, 11, 14, 15, 17, 21, 24, 26, 27, 56) for every participant. At the screening visit, participants will give a medical history and will undergo a physical exam; blood samples will be collected. Participants will undergo pharmacokinetic (PK) sampling which will require that blood be drawn at 0, 1, 2, 6, 12, 24, 48, 72h after the first dose. For multi-dose PK studies, blood samples will be collected at the same time points after the last dose. Participants will undergo pharmacodynamic (PD) sampling which will require that blood be drawn at 0, 6, 12, 24, 48, 72h after the first dose. For steady-state concentration PK and PD studies, blood samples will be collected 5-30 minutes before Chidamide administration on Day 14, 17, 21. If participants agree, their blood samples may be stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Currently receiving cART and having received cART for a minimum of 18 months, HIV-1 plasma RNA <50 copies/mL for at least 1 year (excluding viral load blips)
* CD4 cell count above 350 cells/μL
* Able, willing to give written informed consent and to adhere to therapy and to comply with time requirements for study visits and evaluations
* Adequate vascular access for leukapheresis

Exclusion Criteria:

* Acute HIV-1 infection
* Received blood transfusions or hematopoetic growth factors within 3 months
* Receipt of compounds with HDAC inhibitor-like activity, such as valproic acid within the last 1 month. Potential participants may enroll after a 30-day washout period.
* Any significant acute medical illness in the past 8 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
* Patient has the following laboratory values within 3 weeks before starting the investigational drug

  1. Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  2. Serum total bilirubin ≥1.5 ULN
  3. Serum creatinine levels ≥1.5 x ULN, or calculated creatinine clearance ≤60 ml/min
  4. Platelet count ≤100 x109/L
  5. Absolute neutrophil count ≤1.5x109/L
  6. Serum potassium, magnesium, phosphorus outside normal limits
  7. Total calcium (corrected for serum albumin) or ionized calcium ≤lower normal limits
* A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for Torsades de pointes (e.g. heart failure)
* History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
* History of diabetes mellitus
* Known hypersensitivity to the components of chidamide or its analogues
* Pregnancy or breast feeding, or expecting to father children within the projected duration of the study
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in plasma HIV-1 RNA | Measured on day 0, 1, 2, 3, 8, 11, 14, 15, 17, 21, 24, 25, 26, 27, 56.

SECONDARY OUTCOMES:
Change in cell-associated HIV-1 RNA | Measured on day 0, 1, 2, 3, 11, 21, 24, 26, 56.
Change in cell-associated total HIV-1 DNA | Measured on day 0, 14, 27, 56.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Measured through 56 days after the administration of chidamide.
Change of plasma concentration of chidamide (pharmacokinetic profile) | Measured through 72 hours after the first and last dose of chidamide; 5-30 minutes before chidamide administration on day 14, 17, 21.
  Participants will undergo pharmacokinetic sampling which will require that blood be drawn at 0, 1, 2, 6, 12, 24, 48, 72h after the first and last dose of chidamide and 5-30 minutes before chidamide administration on day 14, 17, 21.
Change of histone acetylation level in CD4+ T cells (pharmacodynamic profile) | Measured through 72 hours after the first dose of chidamide; 5-30 minutes before chidamide administration on day 14, 17, 21.
  Participants will undergo pharmacodynamic sampling which will require that blood be drawn at 0, 6, 12, 24, 48, 72h after the first dose of chidamide and 5-30 minutes before chidamide administration on day 14, 17, 21.

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Sun, M.D., Ph.D., Principal Investigator — Department of Infectious Diseases, Tangdu Hospital, The Fourth Military Medical University
Locations (1):
- Department of Infectious Diseases, Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi, China